CLINICAL TRIAL: NCT03887156
Title: Evaluation of a Donor Testing Kit for the Prediction of Acute GVHD in Patient Receiving a Peripheral Blood Stem Cells Allograft- Predictor 2
Brief Title: Evaluation of a Donor Testing Kit for the Prediction of AGVHD in Patient Receiving a Peripheral Blood Stem Cell Allograft
Acronym: Predictor2
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: SATT (Unknown); SNC Graft Versus Host Disease (Unknown); Imagine Institute (Other); Axonal-Biostatem (Industry); CERBA laboratory (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K180304J
Record Dates: First submitted 2019-03-12; First posted 2019-03-22 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Acute Myeloid Leukemia in Remission; Lymphoma in Remission; Non-progressive Myeloproliferative Syndrome; Myelodysplasia With Stable Blasts is Cell Number and < 10% of Blastocysts; Acute Leukemia Biphenotypic in Remission; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Other): One arm
  Interventions: Diagnostic Test: Ex vivo capacities of CD4neg INkT expansion of the peripheral blood donor with the Predictor test

INTERVENTIONS:
Diagnostic Test: Ex vivo capacities of CD4neg INkT expansion of the peripheral blood donor with the Predictor test — Calculation of ex vivo capacities of CD4neg INkT expansion of the peripheral blood from an identified donor for an allograft. Sample is collected before mobilization and the blood culture and analysis using the Predictor test are performed by the central lab.

SUMMARY:
The aim is to validate an in vitro diagnosis medical device to predict grade II to IV aGVHD after a cell graft

DETAILED DESCRIPTION:
Acute Graft Versus Host Disease (aGVHD) is the most frequent complication in allogeneic Hematopoietic Stem Cell Transplantation (allo-HSCT). It affects up to 50% patients, among whom 15% to 25% develop severe forms, often lethal, yet impossible to predict even for donors with a Human Leukocyte Antigene (HLA) 10/10 compatibility. Global Overall Survival (OS) after transplantation is 40% to 60% only due to post transplant severe complications. There is a major medical need for a technology that would predict the risk of aGVHD and would allow the selection of a favourable donor among multiple Human Leukocyte Antigene (HLA)10/10 compatible donors.

MT. Rubio and M. Bouillié at Pr Olivier Hermine's lab previously reported that enhanced early post-transplant invariant Natural Killer T (iNKT) cells reconstitution from donor cells was correlated to reduced risk of aGVHD, without impairment of the Graft Versus Leukemia (GVL) effect. They subsequently demonstrated that the expansion of donors CD4neg invariant Natural Killer T (iNKT) cells subpopulation was predictive of a reduced risk of aGVHD, and developed a method for predicting this risk based on the expansion factor of CD4neg invariant Natural Killer T (iNKT) cells in the peripheral blood stem cell (PBSC) graft. This invariant Natural Killer T (iNKT) cells functional test reaches its optimal predictive capacity with 94% sensitivity and 100% specificity in allo-HSCT performed with Human Leukocyte Antigene (HLA) 10/10 matched peripheral blood stem cell (PBSC) grafts for non-progressive hematological malignant diseases, in complete response, which represent the majority of the indications of allogeneic HSCT. Similar predictive value was also observed when the test was performed from donor's peripheral blood before G-CSF mobilization. It was not associated with an increased risk of relapse. This test could therefore allow to easily selecting the best donor if different siblings or unrelated donors are available before PBSC allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT :

  * Age between 18 and 65 years ( included )
  * Being candidate to a graft of peripheral hematopoietic stem cells , according the following criteria :
* HLA compatibility 10 / 10 with the selected donor
* Malignant haematological disorder as described below :

  * Acute Myeloid Leukemia (AML) or Acute Lymphoblastic Leukemia ( ALL) in 1st or 2d complete remission
  * Aggressive lymphoma in complete remission
  * Non - progressive myeloproliferative syndrome ,
  * Myelodysplasia with stable blasts is cell number and < 10 % of blastocysts,
  * Acute leukemia biphenotypic in 1st or 2d complete remission
* Sequential graft conditioning, myeloablative or with a reduced intensity, both may include ATG
* Classical scheme for immunosuppression decrease ( from day 90 to day 180 ) • Not being opposed to medical data collection DONOR
* Adult ( ≥ 18 year old) up to the maximum authorized by each National Transplantation Authority
* Being a patient's sibling or registered in the Bone Marrow Donors Worldwide registry or a national registry
* Being candidate to a Peripheral Blood Stem Cells donation with a Human Leucocyt Antigen (HLA) 10 / 10 compatibility with the recipient ,
* Signed and dated informed consent ( in accordance with local regulation of the country in which the observation is performed )

Exclusion Criteria:

* Participating in a clinical trial, if interventional on the prophylaxis treatment ( not on the prophylaxis ) of GVHD, in the 30 days prior to the inclusion and during the Predictor 2 study ,
* Being placed under legal supervision ,
* Presenting any impossibility to fulfil the study requirements, due to geographical, social or physical reasons

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Estimated)
Dates: Start 2019-09-16 (Actual); Primary Completion 2023-03-16 (Estimated); Study Completion 2023-03-16 (Estimated)

PRIMARY OUTCOMES:
Number of aGVHD of grade II to IV observed for the recipients | 3 month after allograft performance
  To predict the risk of acute GVHD. Number of aGVHD of grade II to IV observed for the recipients in the 3 months after the graft and results of the Predictor test, before graft, on their own donor's blood.

SECONDARY OUTCOMES:
Evaluation of medico-economic aspect of the Predictor test Total estimated cost of the aGVHD treatment | 3 month after allograft performance.
  Number of hospitalization or medical consultation, exams, concomitant treatments.
Evaluation of the medico-economic aspect of the Predictor test Total estimated cost of the aGVHD treatment | 3 month after allograft performance.
  Number of medical consultations
Evaluation of the medico-economic aspect of the Predictor test Total estimated cost of the aGVHD treatment | 3 month after allograft performance.
  Number of exams
Evaluation of the medico-economic aspect of the Predictor test Total estimated cost of the aGVHD treatment | 3 month after allograft performance.
  Number of concomitant treatments

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Hermine, MD, Principal Investigator — Head of adult hematology department
Locations (22):
- Belgium (3):
  - Z.N.A. Stuivenberg Ziekenhuis, Antwerp
  - CHU Liège, Liège
  - U.Z. Antwerpen, Wilrijk
- France (16):
  - CHU Amiens-Picardie, Amiens
  - CHU Angers, Angers
  - CHU de Caen, Caen
  - HIA Percy, Clamart
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Dupuyten, Limoges
  - Hôtel Dieu, Nantes
  - CHU Nice, Nice
  - Hôpital de la Pitiè-Salpétrière, Paris
  - Hôpital Necker Enfants Malades, Paris
  - CHU Bordeaux, Pessac
  - CHU de Poitiers, Poitiers
  - CHU de Rennes, Rennes
  - L'Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Institut Universitaire du Cancer de Toulouse, Toulouse
  - CHRU Nancy - Hôpital de Brabois, Vandœuvre-lès-Nancy
- Germany (3):
  - Donor Site - Koln, Cologne
  - Donor Site-Dresden, Dresden
  - Medizinische Hochschule Hannover, Hanover

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rubio MT, Bouillie M, Bouazza N, Coman T, Trebeden-Negre H, Gomez A, Suarez F, Sibon D, Brignier A, Paubelle E, Nguyen-Khoc S, Cavazzana M, Lantz O, Mohty M, Urien S, Hermine O. Pre-transplant donor CD4- invariant NKT cell expansion capacity predicts the occurrence of acute graft-versus-host disease. Leukemia. 2017 Apr;31(4):903-912. doi: 10.1038/leu.2016.281. Epub 2016 Oct 14. PMID 27740636